CLINICAL TRIAL: NCT02127047
Title: Effects of Exercise and Inhibition of Dipeptidyl Peptidase-4 on Insulin Secretion in Subjects With Type 1 Diabetes
Acronym: EXTYPE-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EKBB 349/12
Record Dates: First submitted 2014-04-28; First posted 2014-04-30 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Diabetes Mellitus Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Sitagliptin Phosphate; Exercise

ARMS (2):
- Sitagliptin (Experimental): Patients receive Sitagliptin (100mg/d) without further intervention
  Interventions: Drug: Sitagliptin
- Sitagliptin and exercise (Experimental): Patients receive sitagliptin (100mg/d) and follow a physical training intervention program
  Interventions: Drug: Sitagliptin; Drug: Exercise

INTERVENTIONS:
Drug: Sitagliptin
Drug: Exercise
  Arms: Sitagliptin and exercise

SUMMARY:
Increasing evidence suggests pancreatic islet beta-cell regeneration occurs throughout the course of the disease in patients with type 1 diabetes. Therefore, decreased beta-cell mass in type 1 diabetes may be improved through inhibition of beta-cell destruction and stimulation of proliferation, even after prolonged duration of disease.

Physical activity improves insulin secretion via unknown underlying mechanisms. We recently observed that Interleukin-6 induces glucagon like Peptide (GLP)-1 production and release from the islet alpha-cell and the intestinal L-cell. Furthermore, exercise induces release of Interleukin-6 from skeletal muscle resulting in elevated circulating Interleukin-6 levels. Therefore we hypothesize that exercise-induced Interleukin-6 promotes glucagon like peptide-1 secretion from the islet α-cell and the intestinal L-cell, thereby providing a mechanism how physical activity can help maintain and improve beta-cell function in patients with type 1 diabetes. This mechanism can be enhanced by concomitant dipeptidyl peptidase-IV inhibition.

Physical activity is also known to enhance insulin sensitivity and to attenuate the immune system activity.

Therefore by combining physical activity and dipeptidyl peptidase-IV inhibition we aim to allow for beta-cell regeneration in a interventional randomized open-label study.

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 diabetes (American Diabetes Association criteria) of > 2 year duration that is judged to be stable by the investigator
2. No clinically significant change in treatment regimen for type 1 diabetes (defined as a 20% change) during the 3 months prior to Screening
3. Positive glutamic acid decarboxylase 65 and/or Islet Antigen (IA)-2 auto-antibodies
4. Age ≥ 18 years and ≤ 55 years
5. HbA1c < 7.5% for the previous two measurements including the measurement taken at Screening (both measurements must occur within 6 months prior to enrollment)
6. Body-mass index (BMI) > 18 and < 28 kg/m2
7. Willingness to maintain current doses/regimens of vitamins and dietary supplements through the end of the study
8. For subjects with reproductive potential, a willingness to use contraceptive measures adequate to prevent the subject or the subject's partner from becoming pregnant during the study. Adequate contraceptive measures include hormonal methods used for two or more cycles prior to Screening (e.g., oral contraceptive pills, contraceptive patch, or contraceptive vaginal ring), double barrier methods (e.g., contraceptive sponge, diaphragm used in conjunction with contraceptive foam or jelly, and condom used in conjunction with contraceptive foam or jelly), intrauterine methods (IUD), sterilization (e.g., tubal ligation or a monogamous relationship with a vasectomized partner), and abstinence.

Exclusion Criteria:

1. Regular training of more than 90 minutes / week
2. History or signs of cardiovascular disease, proliferative retinopathy, nephropathy or neuropathy
3. Signs of current infection
4. Neutropenia
5. Anemia
6. Clinically significant kidney or liver disease
7. Current immunosuppressive treatment or documented immunodeficiency

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-11; Primary Completion 2016-07 (Actual); Study Completion 2016-08-05 (Actual)

PRIMARY OUTCOMES:
Change in beta-cell function as derived from change in C-peptide and glucose levels during the mixed meal test | Day 90 compared to baseline (Day 1 pre-dose)

SECONDARY OUTCOMES:
Change in insulin sensitivity as derived from change in C-peptide and glucose levels during the mixed meal test | Day 90 compared to baseline (Day 1 pre-dose)
Change in insulin requirements: 3-day average daily insulin dose | baseline (Day -3 through Day -1) compared to Day 90 (Day 87 through Day 89)
Change in HbA1c levels | baseline (Day 1 pre-dose) at Day 90
Change in fasting glucose | baseline (Day 1 pre-dose) at Day 90
Change in fasting glucagon and cortisol | baseline (Day 1 pre-dose) at Day 90
Change in total number of hypoglycemic events compared to treatment groups | baseline (Day 1 pre-dose) to Day 90
Change in markers of systemic inflammation | from baseline (Day 1 pre-dose) at Day 90
Change in composition of immune cells | from baseline at Day 90
Change in meal-stimulated GLP-1 and gastric inhibitory peptide | Day 90 compared to baseline
Change in lipids profile | baseline at Day 90
Change in fatigue according to the Fatigue Scale for Motor and Cognitive Functions questionnaire | from baseline at Day 90
Change in plasma copeptin and procalcitonin levels | from baseline (Day 1 pre-dose) at Day 90
Change in retinal vascular diameter | Day 90 compared to baseline (Day 1 pre-dose)
Change in arterial stiffness | Day 90 compared to baseline (Day 1 pre-dose)
Change in fractalkine | Day 90 compared to baseline (Day 1 pre-dose)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Donath, Prof. MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland